CLINICAL TRIAL: NCT05483803
Title: CARING: Feasibility Study of Digital Health for Caregivers Emotional and Self-management Support of Children With Type 1 Diabetes
Brief Title: Digital Health Intervention for Caregivers Emotional and Self-management Support of Children With Type 1 Diabetes
Acronym: CARING-T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Hospital Miguel Servet (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CAR-22-001; U1111-1280-9100 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; mhealth; caregiver; emotional health; behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in two sub-studies. Participants in sub-study 1 will be enrolled in an intervention for 1 month. After sub-study 1 completion a new group of participants will be enrolled in the sub-study 2 for the intervention lasting 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualitative sub-study 1 group (Experimental): One group of caregivers (n = 20) will engage with the digital health solution during 1 month.
  Interventions: Behavioral: Adhera® Caring digital intervention for Type 1 Diabetes
- Quantitative sub-study 2 group (Experimental): A different group of caregivers (n = 80) will engage with the digital health solution during 3 months.
  Interventions: Behavioral: Adhera® Caring digital intervention for Type 1 Diabetes

INTERVENTIONS:
Behavioral: Adhera® Caring digital intervention for Type 1 Diabetes — The Adhera® Caring is a mobile based personalized digital intervention for caregivers, lasting for 1 or 3 months (depending on the sub-study).

SUMMARY:
This feasibility study builds upon mental health and technology acceptance theoretical frameworks. It seeks to examine potentials of a mobile-based novel digital health solution based on emotional and behavioral change techniques, to provide emotional and self-management tailored support to caregivers of children with type I diabetes (T1D).

The digital health program, called Adhera® Caring, is designed to be used for approximately 3 months. The study will enroll 100 participants (20 in sub-study 1 and 80 in sub-study 2) who are caregivers of children with type 1 diabetes. There will be a nurse coaching the participants by providing support related to their emotional wellbeing via the mobile solution.

DETAILED DESCRIPTION:
Objectives:

* Primary objective 1. To gather qualitative and quantitative information enabling to better understand psychological burdens that caregivers of children with type 1 diabetes and perceived barriers/facilitators for adoption of a digital health solution.
* Primary objective 2. To assess positive mood states of caregivers of type 1 diabetes patients as an indicator of emotional wellbeing related to the use of the digital health solution.

This is a prospective mixed-methods (qualitative-quantitative) exploratory study composed of two sub-studies:

* Qualitative sub-study 1 (SS1): One group of caregivers (n = 20) will engage with the digital health solution for 1 month. Subsequently, an individual semi-structured interview with each of the participants and a usability questionnaire will proceed to gather user experience qualitative information.
* Quantitative sub-study 2 (SS2): A different group of caregivers (n = 80) will engage with the digital health solution for 3 months. As elaborated in the following sections, a quantitative approach will be adopted to assess different emotional and behavioral parameters before and after engaging with the digital health solution (pre-post design).

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of patients with type 1 diabetes under 18 years of age.
* Patient's debut of type 1 diabetes at least 3 months prior to the start of the study.
* Patients with continuous glucose monitoring.
* Participants with children undergoing insulin treatments (multiple dose insulin or continuous subcutaneous insulin infusion)
* Participants administering insulin treatment to their children
* Users of smartphone whose children are treated with type 1 diabetes treatment for approved indications in Spain.
* Participants must agree on sharing data on continuous glucose monitoring data of their treated children.
* Participants must sign an informed consent
* Participants must be willing to and install the mobile solution of the study.

Exclusion Criteria:

* Candidates without a smartphone or not being able to interact with it.
* Only one legal guardian per child can participate in the study.
* Participants of SS1 will not take part in SS2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Sub-study 1: Qualitative data of psychological burdens experienced as caregivers of children with type 1 diabetes and barriers/facilitators for adopting the digital health solution | 1 Month
  A semi-structured interview based on a mental health and technology acceptance theoretical framework has been specifically designed for this purpose.
Sub-study 2: Changes on caregiver's positive mood | 3 Months
  Positive subscale of the Positive and Negative Affect Scale (PANAS). Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.

SECONDARY OUTCOMES:
Emotional outcome: Changes on caregiver's distress | Baseline up to week 12
  Distress assessed with the depression, anxiety, and stress scale (DASS-21). DASS-21 is a self-report questionnaire consisting of 21 items, 7 items per subscale: depression, anxiety and stress. Patients are asked to score every item on a scale from 0 (did not apply to me at all) to 3 (applied to me very much). Sum scores are computed by adding up the scores on the items per (sub)scale and multiplying them by a factor 2. Sum scores for the total DASS-total scale thus range between 0 and 120, and those for each of the subscales may range between 0 and 42. Cut-off scores of 60 and 21 are used for the total DASS score and for the subscales respectively. Scores ≥60 (for DASS-total) and ≥21 (for the depression subscale) are labeled as "high" or "severe".
Emotional outcome: Changes on caregiver's general wellbeing | Baseline up to week 12
  Assessed with the short form of the Mental Health Continuum - short form questionnaire (MHC-SF). Total sum scores on the MHC-SF can range from 0 to 70, with higher scores indicating higher levels of well-being.
Emotional outcome: Changes on caregiver's perceived self-efficacy | Baseline up to week 12
  Perceived self-efficacy assessment with the General Self-Efficacy Scale (GSE), the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Health-related Quality of Life (HrQoL): Changes on the child's HRQoL | Baseline up to week 12
  Children HRQoL assessment with KIDSCREEN-10 index answered by the caregiver as a proxy. The scores range between 10 and 50, and are linearly converted into 0-100 scale in which higher scores represent better quality of life.
Life-style outcome: Adherence to Mediterranean diet | Baseline up to week 12
  Assessed with the KIDMED questionnaire. This questionnaire consists of 16 questions, where negative answers are scored with 0, while affirmative answers are scored with +1/-1 depending on their positive or negative connotation.
Life-style outcome: physical activity (APALQ) | Baseline up to week 12
  Physical activity assessed with Assessment Physical Activity Levels Questionnaire (APALQ). It is a self-administered questionnaire with 5 items scored 1 to 4/5, in which the sum of the answers classifies the global score in 3 categories: sedentary (5 to 10), moderately active (11-16), very active (+17).
Knowledge of the disease and its treatment. | Baseline up to week 12
  Medical checking questions related to the disease, its treatment and if the patients are following the multiple doses of insulin (MDI) or the continuous subcutaneous insulin infusion (CSII) treatment.
Behavioral outcome: objectively measured children's metabolic control to the treatment | Baseline up to week 12
  Assessed from the sensor used via glucose monitoring
Behavioral outcome: Usability | At week 4 (sub-study 1) or week 12 (sub-study 2)
  mHealth solution usability assessed with the System Usability Scale (SUS) questionnaire. SUS can range between 0 and 100 scores, with higher values representing higher usability.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio de Arriba Muñoz, MD, PhD, Principal Investigator — Unidad de Endocrinología Pediátrica, Hospital Miguel Servet; Luis Fernandez Luque, PhD, Principal Investigator — Adhera Health, Inc.
Locations (1):
- Hospital Miguel Servet, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrasco-Hernandez L, Jodar-Sanchez F, Nunez-Benjumea F, Moreno Conde J, Mesa Gonzalez M, Civit-Balcells A, Hors-Fraile S, Parra-Calderon CL, Bamidis PD, Ortega-Ruiz F. A Mobile Health Solution Complementing Psychopharmacology-Supported Smoking Cessation: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 27;8(4):e17530. doi: 10.2196/17530. PMID 32338624